CLINICAL TRIAL: NCT00243607
Title: Prospective Randomized Feasibility Study on the Self Application of Hydrotherapy to Treat Menopausal Symptoms Caused by Breast Cancer Therapy
Brief Title: Hydrotherapy Against Menopausal Symptoms in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Cornelia von Hagens, Head Complementary & Integrative Medicine, Dep. 4.2, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD175-05
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2009-06

CONDITIONS: Amenorrhea; Hot Flashes
Keywords: climacteric symptoms; breast cancer; hydrotherapy
MeSH Terms: conditions — Amenorrhea; Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate treatment group (SBG) (Experimental): immediate start of hydrotherapy (self treatment) in immediate treatment group (SBG)
  Interventions: Other: hydrotherapy according to Kneipp rules
- waiting group (WG) (No Intervention): start of hydrotherapy (self treatment) after waiting period of 12 weeks

INTERVENTIONS:
Other: hydrotherapy according to Kneipp rules — 2-5 applications of hydrotherapy according to Kneipp rules (self application) per day
  Arms: immediate treatment group (SBG)

SUMMARY:
Breast cancer survivors often suffer from climacteric symptoms caused by treatment or diagnosis of their disease.

Hormone replacement therapy is contraindicated and other pharmacological options may also include the risk of stimulating hormone receptors. Hydrotherapy following the guidelines of naturopathy by S. Kneipp is a non-pharmacological treatment option which may influence climacteric symptoms by affecting the regulation of body temperature. In this study, the regular self application of hydrotherapy after initial training by a professional will be evaluated for its efficacy, practicability, and compatibility.

DETAILED DESCRIPTION:
Patients should use 2-5 different treatment options per day and fulfill a diary for symptoms and adherence to self-treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis
* Menopausal complaints score > 14 (MRS II)
* End of last chemotherapy or radiotherapy > 2 months
* Expected stable disease for the next 6 months

Exclusion Criteria:

* Regular intake of glucocorticoids
* Regular practice of hydrotherapy before inclusion
* Start or change of other treatments/changes of lifestyle in order to influence menopausal symptoms
* Psychiatric disorders with possible influence on compliance and adherence to the protocol
* Other severe or progressive diseases with influence on compliance and adherence to the protocol
* Contraindications to hydrotherapy (severe heart failure, relevant dermatological diseases, Raynaud's Phenomenon [M. Raynaud], peripheral arterial occlusive disease Fontaine stage IIb [VK IIb] or more, acute thrombosis, or thrombophlebitis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Menopausal complaints (MRS II) | 12 and 24 weeks

SECONDARY OUTCOMES:
Cortisol profile (saliva) | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Uehleke, Dr.med. Dr.rer.nat. (PhD), Study Chair — Abt. für Naturheilkunde, Charité-Universitätsmedizin Berlin, Campus Benjamin Franklin, Immanual-Krankenhaus
Locations (1):
- Ambulanz für Naturheilkunde und Integrative Medizin, Heidelberg, Baden-Wurttemberg, Germany